CLINICAL TRIAL: NCT05192759
Title: Effect of Theta-Burst Transcranial Magnetic Stimulation (TBS) for Freezing of Gait
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Anhui Medical University (Other)
Responsible Party: Principal Investigator, WANG KAI, Head, Dept of Neurology & Medical Psychology, Director, Cognitive Neuropsychology Lab, PRC, Anhui Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AHMU-TMS-FOG
Record Dates: First submitted 2022-01-03; First posted 2022-01-14 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Transcranial Magnetic Stimulation; Freezing of Gait
Keywords: Transcranial Magnetic Stimulation; Freezing of gait
MeSH Terms: interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TBS Group (Experimental): Participants will receive active transcranial magnetic stimulation (TMS) daily for 1 week
  Interventions: Device: Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation — The stimulations were performed by MagStim Rapid2.

SUMMARY:
To investigate the treatment effect of Theta-burst Transcranial Magnetic Stimulation (TBS) on patients with freezing of gait (FOG) and the underlying neural mechanism.

DETAILED DESCRIPTION:
This was a open-label clinical trial to assess the efficacy and underlying neural mechanism of TBS among patients with FOG. Forty patients with FOG were treated with TBS for 1 week.

Before the TBS treatment, the Freezing of Gait Questionnaire, the Timed up and go test, the Standing Start 180° Turning Test, the Unified Parkinson's Disease Rating Scale, and the Non-motor Symptom Scale, the Pittsburgh sleep quality index were obtained by a trained investigator to assess baseline severity. The patients had receiving a battery measure of neuropsychological tests(mini-mental state examination, Montreal cognitive assessment, digital span test, verbal fluency test, Hamilton depression/anxiety scale) and magnetic resonance imaging (MRI) scan in multimodalities, electroencephalography (EEG) record and fNIRS.

In the second day after the last treatment, all the tests, MRI 、EEG and fNIRS were reassessed. Patients were instructed to focus their answers on the past 1 week.

The clinical symptom and cognition of participants were followed in one month and two month after the last treatment.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosis of FOG with expertise in movement disorders.
2. the score of item 3 of the FOG questionnaire ≥1.
3. ongoing treatment with a stable dose of any medication for 2 months.
4. 40 years of age or older.

Exclusion Criteria:

1. a history of addiction, psychiatric disorders, or neurological diseases other than PD.
2. focal brain lesions on T1-/T2-weighted fluid-attenuated inversion recovery images.
3. anti-PD medication adjustments during rTMS treatment.
4. history of substance abuse within the past 6 months.
5. nonremovable metal objects in or around the head.
6. previously received rTMS treatment.
7. prior history of seizure or history in first-degree relatives.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-11-22 (Actual); Primary Completion 2028-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
The Standing-Start 180° Turn Test (SS-180) | changes from baseline to 1-week post-treatment
  The participants walk for a distance of five meters from a sitting position and come back to the chair after turning 180° around a traffic cone in a 0.7 m × 0.7 m target box.The time and number of steps during the 180° turn (SS180) are measured.

SECONDARY OUTCOMES:
The timed up and go test (TUG) | changes from baseline to 1-week post-treatment
  The participants walk for a distance of five meters from a sitting position and come back to the chair after turning 180° around a traffic cone in a 0.7 m × 0.7 m target box .The time and number of steps during the whole course are measured.
The Freezing of Gait Questionnaire (FOGQ) | changes from baseline to 1-week post-treatment
  This is an very common clinical motor estimating scale for evaluating FOG symptoms with 6 items and 24' in total. Higher scores indicate worse symptoms.
Unified Parkinson's Disease Rating Scale III (UPDRSIII) | changes from baseline to 1-week post-treatment
  This is an very common clinical motor estimating scale, 14 items and 108' in total. Higher scores indicate worse symptoms.
Non-motor symptoms questionnaire | changes from baseline to 1-week post-treatment
  This is a very common clinical scale with nine domains (30 items). Each item was scored on "severity" range from 1 to 3 and "frequency" range from 1 to 4. Higher scores indicate worse symptoms.
HAMD (Hamilton Depression Scale) | changes from baseline to 1-week post-treatment
  This scale was compiled by Hamilton in 1960, is the most common clinical to assess Depression Scale. In this study, 17 versions were selected, and there were 17 questions. The subjects were assessed for their depression in the past week. Each question scored between 0 and 4 points.Higher scores indicate more depressive symptoms.
HAMA (Hamilton Anxiety Scale) | changes from baseline to 1-week post-treatment
  This scale was compiled by Hamilton in 1959.It was one of the most commonly used scales in psychiatric clinic, including 14 items. It is often used in clinical diagnosis and degree classification of anxiety disorder. The subjects were assessed for their anxiety in the past week. Each question scored between 0 and 4 points. The higher the score, the more symptoms of anxiety.
Pittsburgh sleep quality index (PSQI) | changes from baseline to 1-week post-treatment
  This scale was developed by Dr. Buysse et al., a psychiatrist at the University of Pittsburgh in 1989. The scale is suitable for the evaluation of sleep quality in patients with sleep disorders and mental disorders, as well as for the evaluation of sleep quality in general.Each question scored between 0 and 3 points.The higher the score, the worse sleep quality.

CONTACTS AND LOCATIONS:
Locations (1):
- Cognitive Neuropsychology Lab Anhui Medical University, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yu L, Han J, Chen X, Hu L, Wang M, Zhu M, Cheng J, Liu P, Fang L, Li Y, Wu J, Zhao X, Sun J, Ji GJ, Wang K, Ye R, Hu P. Regional-specific structural and functional changes of posterior cerebellar vermis across different stages of Parkinson's disease with gait dysfunction. NPJ Parkinsons Dis. 2025 Jul 12;11(1):208. doi: 10.1038/s41531-025-01065-1. PMID 40651960